CLINICAL TRIAL: NCT00160784
Title: Arthroscopy and Manipulation vs a Home Therapy Program in the Treatment of Adhesive Capsulitis of the Shoulder - A Prospective Randomized Study
Brief Title: Arthroscopy and Manipulation vs a Home Therapy Program in the Treatment of Adhesive Capsulitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44-1997
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-11

CONDITIONS: Adhesive Capsulitis of the Shoulder
MeSH Terms: conditions — Bursitis | interventions — Arthroscopy; Home Infusion Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopic Manipulation (Active Comparator): Manipulation of Shoulder performed during arthroscopy
  Interventions: Procedure: Arthroscopy; Procedure: Arthroscopic manipulation
- Home exercise program (Active Comparator): Shoulder exercise program performed at home to increase shoulder function
  Interventions: Other: Home therapy

INTERVENTIONS:
Procedure: Arthroscopy — Randomized placement into 2 groups; arthroscopic manipulation or home therapy
  Other Names: No other names
  Arms: Arthroscopic Manipulation
Procedure: Arthroscopic manipulation — Manipulation of shoulder performed during arthroscopy
  Other Names: No other names
  Arms: Arthroscopic Manipulation
Other: Home therapy — Shoulder exercise program performed at home that may increase shoulder function
  Other Names: No other names
  Arms: Home exercise program

SUMMARY:
The purpose of this study is to compare two treatments used for treating frozen shoulder which are arthroscopy and forceful stretching of the shoulder and home stretching therapy to see if one relives pain and improves shoulder motion more quickly. The other purpose is to try and understand what causes frozen shoulder. For this purpose, tissue will be taken from the shoulder during surgery and studied for the presence and level of a protein called cytokine (Connective Tissue Growth Factor)

DETAILED DESCRIPTION:
Adhesive capsulitis of the shoulder is a relatively common entity which is poorly understood and produces a significant amount of morbidity in afflicted patients. The natural history of adhesive capsulitis is only just beginning to be understood. It is a self-limiting disease, but may take 18 to 36 months to resolve. During that time, individuals can suffer a significant amount of pain and miss a large amount of work. Many surgeons have treated this process with early manipulation with the outcome never being reported in a prospective manner. Some authors have advocated conservative non-operative treatment, knowing the natural history in most of these shoulders will be near resolution. The primary purpose of this study is to examine in a prospective randomized manner the results of continuous non-operative management versus arthroscopic capsulectomy. This study will determine if operative intervention with an arthroscopic capsulectomy can shorten the natural history of adhesive capsulitis, and give comparable results with non-operative management at final follow-up of 2 years.

A second purpose of the study is to try and identify the mechanism(s) responsible for adhesive capsulitis. Recent research suggests that cytokines and connective tissue growth factor (CTGF) may be involved in the inflammatory and fibrotic processes. The second purpose of this study involves histological and immunohistochemical analysis of capsular and synovial tissue routinely removed during an arthroscopic capsulectomy. Tissue taken from subjects in the surgical treatment group will be compared to tissue from patients undergoing an arthroscopic capsulectomy for reasons other than adhesive capsulitis (control group). Location and concentration of CTGF will be compared between these groups. If levels of CTGF are elevated in the treatment group as hypothesized, development and testing of agents that specifically reduce the action of CTGF may be indicated. A specific agent blocking CTGF has been developed and is nearing clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* frozen shoulder (pain and stiffness) experienced for at least four months and treatment has not helped.

Exclusion Criteria:

* None

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 1997-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
At the end of two years, the SPADI test, Range of Motion test and Strength test will be used to determine the effect of the intervention. | 2 years

SECONDARY OUTCOMES:
The SPADI, Range of Motion and Strength test will be taken at six weeks, three months, six months, one year and two years to evaluate the condition of the affected shoulder. | 6 wk, 3 mo, 6 mo, 1 yr, 2yr

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Wright, MD, Principal Investigator — University of Florida
Locations (1):
- UF Orthopaedics and Sports Medicine Institute, Gainesville, Florida, United States